CLINICAL TRIAL: NCT01599650
Title: A 24-month, Phase IIIb, Open-label, Randomized, Active Controlled, 3-arm, Multicenter Study Assessing the Efficacy and Safety of an Individualized, Stabilization-criteria-driven PRN Dosing Regimen With 0.5-mg Ranibizumab Intravitreal Injections Applied as Monotherapy or With Adjunctive Laser Photocoagulation in Comparison to Laser Photocoagulation in Patients With Visual Impairment Due to Macular Edema Secondary to Branch Retinal Vein Occlusion
Brief Title: Efficacy and Safety of Ranibizumab With or Without Laser in Comparison to Laser in Branch Retinal Vein Occlusion
Acronym: BRIGHTER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRFB002E2402; 2011-002859-34 (EudraCT Number)
Record Dates: First submitted 2012-05-02; First posted 2012-05-16 (Estimated); Results first posted 2016-11-10 (Estimated); Last update posted 2016-11-10 (Estimated); Status verified 2016-09

CONDITIONS: Branch Retinal Vein Occlusion
Keywords: Macular Edema, Branch Retinal Vein Occlusion, visual impairment
MeSH Terms: conditions — Retinal Vein Occlusion; Macular Edema; Vision Disorders | interventions — Ranibizumab; Lasers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1-ranibizumab monotherapy (Experimental): Ranibizumab 0.5 mg
  Interventions: Drug: Ranibizumab
- 2-ranibizumab with laser (Experimental): Ranibizumab 0.5 mg + laser
  Interventions: Drug: Ranibizumab; Procedure: Laser
- 3-laser monotherapy (Active Comparator): Laser monotherapy with Ranibizumab 0.5 mg from Month 6
  Interventions: Procedure: Laser

INTERVENTIONS:
Drug: Ranibizumab
  Other Names: Lucentis
  Arms: 1-ranibizumab monotherapy; 2-ranibizumab with laser
Procedure: Laser — laser photocoagulation
  Arms: 2-ranibizumab with laser; 3-laser monotherapy

SUMMARY:
This study will generate comparative data for 0.5-mg ranibizumab using PRN dosing administered with or without adjunctive laser treatment versus laser photocoagulation (the current standard of care) up to Month 6 in patients with visual impairment due to ME secondary to BRVO. Additionally the results of this study will provide long-term (24-month) safety and efficacy data for ranibizumab, administered with or without adjunctive laser treatment in this indication.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained before any study assessment is performed
* Diagnosis of visual impairment exclusively due to ME secondary to BRVO
* BCVA score at Screening and Baseline between 73 and 19 letters (ETDRS)

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Stroke or myocardial infarction less than 3 months before Screening
* Uncontrolled blood pressure defined as systolic value of >160 mm Hg or diastolic value of >100 mm Hg at Screening or Baseline.
* Any active periocular or ocular infection or inflammation at Screening or Baseline in either eye
* Uncontrolled glaucoma at Screening or Baseline or diagnosed within 6 months before Baseline in either eye
* Neovascularization of the iris or neovascular glaucoma in the study eye
* Use of any systemic antivascular endothelial growth factor (anti-VEGF) drugs within 6 months before Baseline
* Panretinal laser photocoagulation within 3 months before Baseline or anticipated or scheduled within the next 3 months following Baseline in the study eye
* Focal or grid laser photocoagulation within 4 months before Baseline in the study eye
* Use of intra- or periocular corticosteroids (including sub-Tenon) within 3 months before Screening in the study eye
* Any use of intraocular corticosteroid implants (eg, dexamethasone [Ozurdex®], fluocinolone acetonide [Iluvien®]) in the study eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 455 (Actual)
Dates: Start 2012-05; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (74):
- Australia (4):
  - Novartis Investigative Site, Parramatta, New South Wales
  - Novartis Investigative Site, Sydney, New South Wales
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Canada (7):
  - Novartis Investigative Site, Calgary, Alberta
  - Novartis Investigative Site, Vancouver, British Columbia
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Halifax, Nova Scotia
  - Novartis Investigative Site, London, Ontario
  - Novartis Investigative Site, Boisbriand, Quebec
  - Novartis Investigative Site, Montreal, Quebec
- Czechia (2):
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
- Novartis Investigative Site, Glostrup Municipality, Denmark
- France (4):
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Lyon
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
- Greece (6):
  - Novartis Investigative Site, Pátrai, Greece
  - Novartis Investigative Site, Thessaloniki, Greece
  - Novartis Investigative Site, Athens, GR
  - Novartis Investigative Site, Heraklion Crete, GR
  - Novartis Investigative Site, Larissa, GR
  - Novartis Investigative Site, Thessaloniki, GR
- Hungary (2):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
- Ireland (2):
  - Novartis Investigative Site, Dublin, Ireland
  - Novartis Investigative Site, Dublin
- Italy (7):
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Milan, MI
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Torino, TO
  - Novartis Investigative Site, Bari
  - Novartis Investigative Site, Udine
- Netherlands (3):
  - Novartis Investigative Site, Leiden 2333 ZA, Netherlands
  - Novartis Investigative Site, Rotterdam
  - Novartis Investigative Site, Tilburg
- Poland (6):
  - Novartis Investigative Site, Bielsko-Biala
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Krakow
  - Novartis Investigative Site, Lublin
  - Novartis Investigative Site, Warsaw
  - Novartis Investigative Site, Wroclaw
- Portugal (4):
  - Novartis Investigative Site, Porto, Porto District
  - Novartis Investigative Site, Coimbra, Portugal
  - Novartis Investigative Site, Porto, Portugal
  - Novartis Investigative Site, Lisbon
- Slovakia (4):
  - Novartis Investigative Site, Žilina, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Banská Bystrica
  - Novartis Investigative Site, Bratislava
- Spain (8):
  - Novartis Investigative Site, Bilbao, Basque Country
  - Novartis Investigative Site, Valladolid, Castille and León
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, L'Hospitalet de Llobregat, Catalonia
  - Novartis Investigative Site, Santiago de Compostela, Galicia
  - Novartis Investigative Site, Madrid, Madrid
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
- Novartis Investigative Site, Örebro, Sweden
- Switzerland (4):
  - Novartis Investigative Site, Olten, Switzerland
  - Novartis Investigative Site, Zurich, Switzerland
  - Novartis Investigative Site, Bern
  - Novartis Investigative Site, Lausanne
- United Kingdom (9):
  - Novartis Investigative Site, Frimley, Surrey
  - Novartis Investigative Site, London, United Kingdom
  - Novartis Investigative Site, Belfast
  - Novartis Investigative Site, Birmingham
  - Novartis Investigative Site, Bristol
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Plymouth
  - Novartis Investigative Site, Southampton

REFERENCES:
- [Derived] Pawloff M, Bogunovic H, Gruber A, Michl M, Riedl S, Schmidt-Erfurth U. SYSTEMATIC CORRELATION OF CENTRAL SUBFIELD THICKNESS WITH RETINAL FLUID VOLUMES QUANTIFIED BY DEEP LEARNING IN THE MAJOR EXUDATIVE MACULAR DISEASES. Retina. 2022 May 1;42(5):831-841. doi: 10.1097/IAE.0000000000003385. PMID 34934034
- [Derived] Tadayoni R, Waldstein SM, Boscia F, Gerding H, Gekkieva M, Barnes E, Das Gupta A, Wenzel A, Pearce I; BRIGHTER Study Group. Sustained Benefits of Ranibizumab with or without Laser in Branch Retinal Vein Occlusion: 24-Month Results of the BRIGHTER Study. Ophthalmology. 2017 Dec;124(12):1778-1787. doi: 10.1016/j.ophtha.2017.06.027. Epub 2017 Aug 12. PMID 28807635
- [Derived] Tadayoni R, Waldstein SM, Boscia F, Gerding H, Pearce I, Priglinger S, Wenzel A, Barnes E, Gekkieva M, Pilz S, Mones J; BRIGHTER study group. Individualized Stabilization Criteria-Driven Ranibizumab versus Laser in Branch Retinal Vein Occlusion: Six-Month Results of BRIGHTER. Ophthalmology. 2016 Jun;123(6):1332-44. doi: 10.1016/j.ophtha.2016.02.030. Epub 2016 Mar 30. PMID 27039022

RESULTS

PARTICIPANT FLOW:
Groups:
- 1-ranibizumab Monotherapy: laser therapy + Ranibizumab 0.5 mg
- 3-laser Monotherapy: after 6 months, laser patients could be treated with ranibizumab
Period: Overall Study
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Started | 183 | 180 | 92
Completed 6 Mos | 174 | 170 | 80
Completed | 161 | 154 | 65
Not Completed | 22 | 26 | 27
Not completed — Administrative issue | 1 | 0 | 1
Not completed — Physician Decision | 2 | 0 | 7
Not completed — Protocol Violation | 0 | 3 | 0
Not completed — Death | 2 | 1 | 2
Not completed — Lost to Follow-up | 3 | 3 | 3
Not completed — Withdrawal by Subject | 11 | 11 | 10
Not completed — Adverse Event | 3 | 8 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy | Total
Number analyzed (Participants) | 183 | 180 | 92 | 455
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.7 (10.34) | 67.3 (10.41) | 67.7 (9.67) | 66.3 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 90 | 84 | 55 | 229
  Male | 93 | 96 | 37 | 226

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Visual Acuity: BCVA Change at Month 6 Compared to Baseline in Patients With Visual Impairment Due to Branch Retinal Vein Occlusion (BRVO)
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)
  -like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. For the mean change of best corrected visual acuity at Month 6 compare to Baseline, the 95% confidence interval and P value (related to the null hypothesis that this mean change is equal to zero) based on a t distribution/t test were calculated and assessed by an ANOVA model.
Time Frame: Baseline, 6 Months
Population: analysis for change consists of the group that had a baseline and 6 month data point
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
letters
  Baseline | 59.5 (11.78) | 56.6 (13.19) | 56.8 (13.86)
  Month 6 | 74.3 (12.27) | 71.4 (14.43) | 62.8 (14.08)
  Change from Baseline atMonth 6 | 14.8 (10.70) | 14.8 (11.13) | 6.0 (14.27)
Statistical Analysis 1: Comparison: 1-ranibizumab Monotherapy vs 3-laser Monotherapy; Test type: Superiority or Other; p < 0.0001, ANOVA; difference in LS mean = 10.0, 95% CI 2-sided [7.3 to 12.8], Standard Error of Mean 1.41
Statistical Analysis 2: Comparison: 2-ranibizumab With Laser vs 3-laser Monotherapy; Test type: Superiority or Other; p < 0.0001, ANOVA; difference in LS Means = 8.7, 95% CI 2-sided [5.8 to 11.6], Standard Error of Mean 1.46

2. Secondary Outcome: The Mean Average Change in Visual Acuity From Month 1 Through Month 24 Compared to Baseline
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. (A positive average change from baseline of BCVA indicates improvement): Mean Average Change: for each patient, first average change is calculated as the average of the changes from baseline to Month 1 over Month 24. Then, mean average change is calculated as the average of average changes across all patients.
Time Frame: Baseline, 24 Months
Population: analysis for change consists of the group that had a baseline and 24 month data point
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
letters
  Baseline | 59.5 (11.78) | 56.6 (13.19) | 56.8 (13.86)
  Average Month 1 toMonth 24 | 74.5 (12.11) | 72.0 (13.56) | 65.9 (13.24)
  Change from Baseline | 15.0 (10.86) | 15.4 (10.76) | 9.1 (13.49)

3. Secondary Outcome: Number of Ranibizumab Treatments From Day 1 to Month 23 by Treatment Group
Description: Number of injections provided to the patients during the 23 month period and conducted within FAS with LOCF and observed data.
Time Frame: Day 1 through Month 23
Measure: Mean (Standard Deviation); unit: treatments
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser
Number analyzed (Participants) | 180 | 178
treatments | 11.4 (5.76) | 11.3 (6.03)

4. Secondary Outcome: Mean Average Change in Visual Acuity (BCVA Letters) From Month 1 Through Month 6
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) -like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters.(A positive average change from baseline of BCVA indicates improvement): Mean Average Change: for each patient, first average change is calculated as the average of the changes from baseline to Month 1 over Month 6. Then, mean average change is calculated as the average of average changes across all patients.
Time Frame: From Baseline through Month 6
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
letters
  Baseline | 59.5 (11.78) | 56.6 (13.19) | 56.8 (13.86)
  Average Month 1 to Month 6 | 72.7 (11.49) | 69.7 (13.38) | 61.7 (12.66)
  Change from Baseline | 13.2 (9.60) | 13.2 (9.89) | 4.8 (11.69)

5. Secondary Outcome: The Mean Change in Visual Acuity BCVA (Letters) From Baseline at Month 12 and Month 24
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS) -like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. For the mean change of best corrected visual acuity at Month 12 and Month 24 compare to Baseline, the 95% confidence interval and P value (related to the null hypothesis that this mean change is equal to zero) based on a t distribution/t test were calculated and were assessed by an ANOVA model.
Time Frame: Baseline, Month 12 and Month 24
Population: Full Analysis set
Measure: Mean (Standard Deviation); unit: letters
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
letters
  Baseline | 59.5 (11.78) | 56.6 (13.19) | 56.8 (13.86)
  Month 12 | 74.9 (12.87) | 72.3 (15.31) | 66.8 (13.87)
  Change from baseline Month 12 | 15.4 (12.25) | 15.7 (13.12) | 10.0 (14.33)
  Month 24 | 75.0 (14.65) | 73.9 (14.59) | 68.4 (15.26)
  Change from baseline Month 24 | 15.5 (13.91) | 17.3 (12.61) | 11.6 (16.09)

6. Secondary Outcome: The Percent of Patients With a Visual Acuity Gain of ≥1, ≥5, ≥10, ≥15, and ≥30 Letters From Baseline up to Month 6 and Month 24, by Visit
Description: BCVA score was based on the number of letters read correctly on the Early Treatment Diabetic retinopathy Study (ETDRS) visual acuity chart assessed at a starting distance of 4 meters. An increased score indicates improvement in acuity. This outcome assessed the number of participants who had improvement of ≥1, ≥5, ≥10, ≥15, and ≥30 letters of visual acuity at Month 6 & Month 24 as compared with baseline, was assessed by an ANOVA model. Endpoints related to the proportion of patients with BCVA letter gain or loss from Baseline was analyzed via stratified Cochran-Mantel-Haenszel test with stratification based on baseline BCVA (baseline BCVA less than or equal to 39, 40 to 59, greater than or equal to 60 letters, treatment groups).
Time Frame: Baseline, Month 6 and Month 24
Measure: Number; unit: percent patients gaining improvement
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
percent patients gaining improvement
  BCVA improvement of >= 1 lettermonth 6 | 93.3 | 96.1 | 63.3
  BCVA improvement of >= 1 lettermonth 24 | 89.4 | 93.8 | 77.8
  BCVA improvement of >= 5 lettersmonth 6 | 86.1 | 88.2 | 50.0
  BCVA improvement of >= 5 lettersmonth 24 | 83.3 | 89.3 | 70.0
  BCVA improvement of >= 10 lettersmonth 6 | 66.7 | 68.5 | 41.1
  BCVA improvement of >= 10 lettersmonth 24 | 71.1 | 75.8 | 60.0
  BCVA improvement of >= 15 lettersmonth 6 | 45.0 | 47.2 | 27.8
  BCVA improvement of >= 15 lettersmonth 24 | 52.8 | 59.6 | 43.3
  BCVA improvement of >= 30 lettersmonth 6 | 10.0 | 9.6 | 3.3
  BCVA improvement of >= 30 lettersmonth 24 | 13.3 | 14.0 | 11.1

7. Secondary Outcome: Number of Patients With a BCVA Improvement vs Baseline or Achieving Greater Than or Equal to 73 Letters at Month 6 in the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart at baseline and Month 6 while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. BCVA above 73 letters at Month 6 indicates a positive outcome.
Time Frame: Month 6
Measure: Number; unit: participants
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
participants
  BCVA improvement of ≥ 1 letter | 168 | 171 | 57
  BCVA improvement of ≥ 5 letters N | 155 | 157 | 45
  BCVA improvement of ≥ 10 letters | 120 | 122 | 37
  BCVA improvement of ≥ 15 letters | 81 | 84 | 25
  BCVA improvement of ≥ 30 letters | 18 | 17 | 3
  BCVA score ≥ 73 letters | 118 | 97 | 28

8. Secondary Outcome: Number of Patients With a BCVA Improvement vs Baseline or Achieved Greater Than or Equal to 73 Letters at Month 24 in the Study Eye
Description: Best Corrected Visual Acuity (BCVA) was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)-like chart at baseline and Month 12 while participants were in a sitting position at a testing distance of 4 meters. The range of EDTRS is 0 to 100 letters. BCVA above 73 letters at Month 24 indicates a positive outcome.
Time Frame: Month 24
Measure: Number; unit: participants
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
participants
  BCVA improvement of ≥ 1 letter | 161 | 167 | 70
  BCVA improvement of ≥ 5 letters | 150 | 159 | 63
  BCVA improvement of ≥ 10 letters | 129 | 135 | 54
  BCVA improvement of ≥ 15 letters | 95 | 106 | 39
  BCVA improvement of ≥ 30 letters | 24 | 25 | 10
  BCVA score ≥ 73 letters | 119 | 114 | 41

9. Secondary Outcome: The Mean Change in Central Reading Center-assessed Central Subfield Thickness From Month 12 and Month 24 vs. Baseline by Treatment Arm
Description: Retinal thickness was measured using Optical Coherence Tomography (OCT). The images were reviewed by a central reading center to ensure a standardized evaluation. Stratification was done based on categories of baseline best corrected visual acuity & analysis was based on analysis of variance (ANOVA)
Time Frame: Month 12 and Month 24
Measure: Mean (Standard Error); unit: microns
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
microns
  month 12 | -215.9 (12.83) | -242.5 (14.14) | -203.9 (22.22)
  month 24 | -228.1 (12.65) | -261.7 (15.20) | -232.7 (24.38)

10. Secondary Outcome: The Mean Change in Patient Reported Outcomes in NEI-VFQ-25 Score (Composite Score and Subscales) at Month 6 and Month 24 Compared to Baseline
Description: The survey consists of 25 items representing 11 vision related constructs (general vision, ocular pain, near activities, distance activities, social functioning, mental health, role difficulties, dependency, driving, color vision, peripheral vision) plus a single-item general health rating question. All items are scored so that a high score represents better functioning. Each item is then converted to a 0 to 100 scale so that the lowest and highest possible scores are set at 0 and 100 points, respectively. In this format scores represent the achieved percentage of the total possible score, e.g. a score of 50 represents 50% of the highest possible score.
Time Frame: Months 6 and 24
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 1-ranibizumab Monotherapy | 2-ranibizumab With Laser | 3-laser Monotherapy
Number analyzed (Participants) | 180 | 178 | 90
score on a scale
  month 6 composite score | 5.6 (9.56) | 4.2 (10.41) | 3.7 (12.12)
  month 24 composite score | 8.0 (11.78) | 5.0 (11.44) | 4.9 (14.79)

11. Secondary Outcome: BCVA (Letters) Mean Average Change From First Ranibizumab Treatment to Month 24 in the Study Eye for Patients Randomized to the Laser Monotherapy Arm
Description: Best-Corrected Visual Acuity (BCVA) letters was measured using Early Treatment Diabetic Retinopathy Study (ETDRS)
  -like chart while participants were in a sitting position at a testing distance of 4 meters. The range of ETDRS is 0 to 100 letters. For the mean change of best corrected visual acuity at Month 24 compare to Baseline, the 95% confidence interval and P value (related to the null hypothesis that this mean change is equal to zero) based on a t distribution/t test were calculated and assessed by an ANOVA model.
Time Frame: Month 24
Population: Randomized set
Measure: Mean (Standard Deviation); unit: BCVA letters
Groups:
- 3- Laser Monotherapy: laser therapy + Ranibizumab 0.5 mg after Month 6
Arm/Group | 3- Laser Monotherapy
Number analyzed (Participants) | 66
BCVA letters
  Value at 1st Ranibizumab treatment | 61.7 (12.21)
  Average post 1st treatment through Month 24 | 68.16 (11.84)
  Change from 1st Ranibizumab treatment | 6.49 (7.83)

ADVERSE EVENTS:
Time Frame: [1] Safety set was summarized based on actual treatment received. There were 3 laser monotherapy patients who received ranibizumab and 1 ranibizumab patient who received laser treatment which resulted in percentages > 100% for the ranibizumab + laser arm.
Groups:
- Ranibizumab 0.5mg: Ranibizumab 0.5mg
- Ranibizumab 0.5mg + Laser: Ranibizumab 0.5mg + Laser
  [1] Safety set was summarized based on actual treatment received. There were 3 laser monotherapy patients who received ranibizumab and 1 ranibizumab patient who received laser treatment which resulted in percentages > 100% for the ranibizumab + laser arm.
- Laser Monotherapy With Ranibizumab 0.5 mg From Month 6: Laser monotherapy with Ranibizumab 0.5 mg from Month 6
- Laser Monotherapy Without Ranibizumab 0.5 mg From Month 6: Laser monotherapy without Ranibizumab 0.5 mg from Month 6
Arm/Group | Ranibizumab 0.5mg | Ranibizumab 0.5mg + Laser | Laser Monotherapy With Ranibizumab 0.5 mg From Month 6 | Laser Monotherapy Without Ranibizumab 0.5 mg From Month 6
Serious Adverse Events (participants affected / at risk) | 30/180 | 33/183 | 10/63 | 3/25
Other Adverse Events (participants affected / at risk) | 112/180 | 121/183 | 40/63 | 14/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=180) | Ranibizumab 0.5mg + Laser (N=183) | Laser Monotherapy With Ranibizumab 0.5 mg From Month 6 (N=63) | Laser Monotherapy Without Ranibizumab 0.5 mg From Month 6 (N=25)
Acute coronary syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0
Aortic valve incompetence (Cardiac disorders) | 1 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 1 | 0
Arteriosclerosis coronary artery (Cardiac disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 3 | 1 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 1 | 0 | 0
Coronary artery embolism (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Cataract (Fellow untreated eye) (Eye disorders) | 1 | 0 | 0 | 0
Cataract (Study eye) (Eye disorders) | 1 | 0 | 0 | 0
Macular fibrosis (Study eye) (Eye disorders) | 0 | 0 | 1 | 0
Macular hole (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Retinal aneurysm (Fellow untreated eye) (Eye disorders) | 0 | 1 | 0 | 0
Retinopathy (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 1 | 1 | 0 | 0
Vitreous haemorrhage (Study eye) (Eye disorders) | 0 | 1 | 0 | 0
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Intestinal polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 2 | 0 | 0
Gallbladder disorder (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatic mass (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Dengue fever (Infections and infestations) | 0 | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Perichondritis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0 | 0
Facial bones fracture (Fellow untreated eye) (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Periprosthetic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Intraocular pressure increased (Fellow untreated eye) (Investigations) | 0 | 1 | 0 | 0
Intraocular pressure increased (Study eye) (Investigations) | 0 | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0
Basal ganglia stroke (Nervous system disorders) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Burnout syndrome (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal failure chronic (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dermatitis bullous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0
Hypovolaemic shock (Vascular disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ranibizumab 0.5mg (N=180) | Ranibizumab 0.5mg + Laser (N=183) | Laser Monotherapy With Ranibizumab 0.5 mg From Month 6 (N=63) | Laser Monotherapy Without Ranibizumab 0.5 mg From Month 6 (N=25)
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 2 | 0
Blepharitis (Fellow untreated eye) (Eye disorders) | 2 | 11 | 0 | 0
Blepharitis (Study eye) (Eye disorders) | 3 | 11 | 1 | 0
Cataract (Fellow untreated eye) (Eye disorders) | 3 | 6 | 0 | 0
Cataract (Study eye) (Eye disorders) | 8 | 3 | 1 | 0
Conjunctival haemorrhage (Study eye) (Eye disorders) | 15 | 15 | 5 | 0
Conjunctivitis allergic (Study eye) (Eye disorders) | 5 | 1 | 0 | 0
Corneal erosion (Study eye) (Eye disorders) | 0 | 4 | 0 | 0
Cystoid macular oedema (Study eye) (Eye disorders) | 4 | 1 | 1 | 0
Dry eye (Fellow untreated eye) (Eye disorders) | 9 | 3 | 2 | 0
Dry eye (Study eye) (Eye disorders) | 10 | 3 | 2 | 0
Eye irritation (Study eye) (Eye disorders) | 4 | 7 | 1 | 0
Eye pain (Study eye) (Eye disorders) | 18 | 21 | 3 | 0
Eye pruritus (Study eye) (Eye disorders) | 4 | 2 | 2 | 0
Eyelid oedema (Study eye) (Eye disorders) | 4 | 3 | 0 | 0
Glaucoma (Study eye) (Eye disorders) | 4 | 2 | 0 | 0
Lacrimation increased (Study eye) (Eye disorders) | 5 | 2 | 1 | 0
Macular fibrosis (Study eye) (Eye disorders) | 8 | 7 | 1 | 0
Macular oedema (Study eye) (Eye disorders) | 4 | 5 | 3 | 1
Metamorphopsia (Study eye) (Eye disorders) | 1 | 0 | 2 | 0
Ocular hyperaemia (Study eye) (Eye disorders) | 7 | 8 | 0 | 0
Ocular hypertension (Fellow untreated eye) (Eye disorders) | 3 | 4 | 1 | 1
Ocular hypertension (Study eye) (Eye disorders) | 5 | 4 | 0 | 2
Photopsia (Study eye) (Eye disorders) | 2 | 2 | 2 | 0
Posterior capsule opacification (Study eye) (Eye disorders) | 2 | 0 | 2 | 0
Punctate keratitis (Study eye) (Eye disorders) | 6 | 1 | 1 | 0
Retinal haemorrhage (Study eye) (Eye disorders) | 5 | 3 | 2 | 1
Retinal ischaemia (Study eye) (Eye disorders) | 2 | 4 | 1 | 0
Retinal neovascularisation (Study eye) (Eye disorders) | 2 | 1 | 1 | 1
Retinal vein occlusion (Study eye) (Eye disorders) | 0 | 1 | 0 | 1
Vision blurred (Study eye) (Eye disorders) | 1 | 6 | 0 | 0
Visual acuity reduced (Study eye) (Eye disorders) | 5 | 6 | 4 | 1
Vitreous adhesions (Study eye) (Eye disorders) | 1 | 2 | 2 | 0
Vitreous detachment (Study eye) (Eye disorders) | 8 | 7 | 1 | 0
Vitreous floaters (Study eye) (Eye disorders) | 7 | 10 | 4 | 1
Vitreous haemorrhage (Study eye) (Eye disorders) | 5 | 6 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 2 | 3 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 8 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 2 | 2 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 2 | 2 | 0
Oedema peripheral (General disorders) | 6 | 2 | 2 | 0
Acute sinusitis (Infections and infestations) | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 3 | 1 | 1 | 1
Conjunctivitis (Fellow untreated eye) (Infections and infestations) | 1 | 5 | 1 | 0
Conjunctivitis (Study eye) (Infections and infestations) | 1 | 4 | 1 | 0
Herpes zoster (Infections and infestations) | 2 | 4 | 1 | 0
Influenza (Infections and infestations) | 13 | 13 | 2 | 1
Laryngitis (Infections and infestations) | 2 | 0 | 1 | 1
Nasopharyngitis (Infections and infestations) | 15 | 17 | 4 | 1
Onychomycosis (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 4 | 2 | 1 | 0
Sinusitis (Infections and infestations) | 8 | 2 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 6 | 6 | 3 | 0
Urinary tract infection (Infections and infestations) | 6 | 4 | 3 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 1 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 6 | 3 | 0
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Procedural pain (Injury, poisoning and procedural complications) | 4 | 1 | 0 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood pressure increased (Investigations) | 3 | 0 | 0 | 1
Intraocular pressure increased (Study eye) (Investigations) | 17 | 17 | 2 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 3 | 3 | 2 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 3 | 6 | 0 | 0
Hyperlipidaemia (Metabolism and nutrition disorders) | 2 | 0 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 2 | 2 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 1 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 5 | 8 | 3 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 7 | 0 | 0
Dizziness (Nervous system disorders) | 2 | 6 | 0 | 1
Headache (Nervous system disorders) | 11 | 9 | 6 | 0
Migraine (Nervous system disorders) | 0 | 4 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 1
Sciatica (Nervous system disorders) | 0 | 0 | 2 | 0
Visual field defect (Fellow untreated eye) (Nervous system disorders) | 0 | 0 | 0 | 1
Depression (Psychiatric disorders) | 1 | 4 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 6 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0 | 0
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 19 | 22 | 7 | 2
Phlebitis superficial (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.